CLINICAL TRIAL: NCT01244074
Title: Visual Rehabilitation of Patients With Myopic Maculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Other Study IDs: BIO0210
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-02

CONDITIONS: Myopic Maculopathy

ARMS (1):
- biofeedback (Experimental)
  Interventions: Behavioral: biofeedback training

INTERVENTIONS:
Behavioral: biofeedback training

SUMMARY:
The Visual Pathfinder (LACE inc.) offers a non- invasive, patient- centered visual rehabilitation system based on an acoustic biofeedback. The investigators wanted to evaluate its usefulness in the improvement of visual function in visually impaired patients with high myopia.

ELIGIBILITY:
Inclusion Criteria:

* high myopia (range 9-15 D) visited at the Outpatient Medical Retina's Hospital A. Fiorini Terracina (LT), University of Rome "La Sapienza", Polo Pontino. The diagnosis of myopic maculopathy was made on the basis of a comprehensive ophthalmological evaluation which included: biomicroscopic examination of anterior and posterior segment, fluorescein angiography (FAG) (Heidelberg HRA-2, FA module Heidelberg, Germany), optical coherence tomography (OCT), Spectral Domain (Heidelberg HRA-2, OCT module Heidelberg, Germany) and microperimetry with microperimeter MP-1 (Nidek Technologies, Padova, Italy).

Exclusion Criteria:

* The investigators have excluded patients with other eye diseases (glaucoma, AMD, retinal detachment, etc.), uncooperative patients and persons with opacity of the dioptric media.

Ages: 35 Years to 57 Years | Sex: All
Age Groups: Adult

PRIMARY OUTCOMES:
improvement of visual performance

SECONDARY OUTCOMES:
improvement of visual acuity, retinal sensitivity, fixation stability

CONTACTS AND LOCATIONS:
Locations (1):
- University La Sapienza, Polo Pontino, Latina, Italy